CLINICAL TRIAL: NCT03654807
Title: The Effect of High Intensity Walking on Frailty
Brief Title: The Effect of Walking on Frailty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Margaret Danilovich, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00207757
Record Dates: First submitted 2018-08-21; First posted 2018-08-31 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Walking (Experimental): HIW (70-80% HRmax)
  Interventions: Behavioral: High Intensity Walking
- Casual Speed Walking (Experimental): Self selected pace
  Interventions: Behavioral: Casual Speed Walking

INTERVENTIONS:
Behavioral: High Intensity Walking — 70-80% HRmax
  Arms: High Intensity Walking
Behavioral: Casual Speed Walking — Self selected pace
  Arms: Casual Speed Walking

SUMMARY:
The purpose of this study is to test the effect of walking intensity on both frailty category (i.e., frail, pre-frail, and nonfrail) and frailty score as a continuous outcome on the SHARE-FI (frailty instrument). As well as test the effect of walking intensity on mobility, physical function, balance, and total Physical Activity.

DETAILED DESCRIPTION:
Frailty impacts up to 60% of older adults and is a leading cause of dependency among older adults. Frail older adults experience physical problems such as balance difficulties, weakness, decreased endurance, and reduced walking speed that increase risk for falls, hospitalizations, institutionalization, and death. Physical activity has multi-system health benefits and is the most recommended frailty management intervention, but guidelines regarding the specific intensity of physical activity remain unclear. High intensity physical activity is an established and safe therapeutic approach in other populations, but it is unclear as to the extent to which high intensity activity can reduce or reverse frailty. This cluster-randomized study will compare a high intensity walking (HIW) intervention to a self-selected, casual speed walking (CSW) intervention implemented within retirement communities for pre-frail and frail older adults. Investigators will randomize 10 retirement communities with 20 participants at each site (200 total participants) to either a 4-month HIW or CSW intervention. All participants will receive 48, individually supervised overground walking sessions occurring within their retirement community. At the beginning and end of the study, investigators will measure participants' frailty, mobility, physical functioning, balance, and total physical activity measured via an ActivPal accelerometer worn for a 1-week observation period to compare which treatment strategy, HIW or CSW, worked better to reduce frailty (aim #1). Investigators will use the SHARE-Frailty Instrument to evaluate frailty as both a categorical (e.g. non-frail, pre-frail, or frail) and a continuous outcome. This approach will allow investigators to determine how participants move between frailty categories as well as within frailty categories in response to intervention. In aim #2, investigators will determine the effect of walking intensity on mobility, physical functioning, balance, and total physical activity. Investigators hypothesize that HIW participants will show decreased frailty and improved mobility, physical functioning, balance, and physical activity at 4 months. Currently, the optimal physical activity guidelines for older adults with frailty are uncertain. Results from this study will provide important knowledge to inform activity guidelines for older adults with frailty and information on a transformative approach to reducing frailty, improving function, and increasing physical activity among a growing segment of the older adults population.

ELIGIBILITY:
Inclusion Criteria:

* • > 60 years of age with pre-frailty or frailty as determined on the SHARE-FI.

  * Able to ambulate at least 10 feet with moderate assistance (<50% physical assistance) or less. Participants will be able to use their assistive device (e.g. cane or walker) during sessions.
  * Resident of one of the 10 enrolled retirement community locations. Individuals must be > 60 years of age to move into the retirement communities by virtue of the individual community policies.
  * Provision of informed consent and clearance for participation as determined by the Exercise and Screening for You (EASY).

Exclusion Criteria:

* • Uncontrolled cardiovascular, metabolic, renal, or respiratory disease that limits exercise participation (e.g., previous heart attack within 3 months of enrollment or uncontrolled diabetes)

  * Resting blood pressure > 180/110 mmHg.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Change in frailty as measured by the Survey of Health, Ageing, and Retirement in Europe-Frailty Instrument (SHARE-FI) | Baseline and four months
  SHARE-FI which assesses fatigue, appetite, weakness, walking difficulties, and low physical activity

SECONDARY OUTCOMES:
Improved mobility as measured by gait speed | Baseline and four months
  Measures related to overall health and mobility
Improved physical function on the Short Physical Performance Battery | Baseline and four months
  Provide an overall assessment of functional status and physical performance
Improved balance as measured by the Berg Balance Scale | Baseline and four months
  The Berg Balance Scale is a valid and reliable 14 item tool to evaluate static and dynamic balance among older adults. Minimum Score 0 to Maximum Score 56. • Score of < 45 indicates individuals may be at greater risk of falling
Total daily physical activity | Baseline and Four Months
  ActivPal Activity Monitors worn for a one week ambulatory monitoring period, data are sampled at 20 Hz in 10 second intervals.
Improved mobility as measured by Time Up and Go | Baseline and Four Months
  Measures related to mobility
Improved mobility as measured by 6 Minute Walk Test | Baseline and Four Months
  Measures related to mobility
Improved balance as measured by the Falls Efficacy | Baseline and Four Months
  Falls Efficacy Scale as this is a widely-used measure among older adults that evaluates the fear of falling and balance confidence, 10-item questionnaire with scores ranging from minimum score 0 to maximum score 100. A total score of greater than 70 indicates that the person has a fear of falling

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Danilovich, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Univiersity Department of Physical Therapy and Human Movement Sciences, Chicago, Illinois, United States

REFERENCES:
- [Derived] Davila VS, Conroy DE, Danilovich MK. Factors That Influence Walking Intervention Adherence for Older Adults Living in Retirement Communities. J Aging Phys Act. 2022 Feb 1;30(1):65-72. doi: 10.1123/japa.2020-0279. Epub 2021 Aug 12. PMID 34384049